CLINICAL TRIAL: NCT01439867
Title: An Open-label, Single-arm Study to Assess the Safety & Tolerability of Cinacalcet in Addition to Standard of Care in Pediatric Subjects Age 28 Days to < 6 Yrs With Chronic Kidney Disease & Secondary Hyperparathyroidism Receiving Dialysis
Brief Title: Safety & Tolerability of Cinacalcet in Pediatric Patients With Chronic Kidney Disease and Secondary Hyperparathyroidism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Amgen decided to terminate the study early to be able to meet US regulatory timelines fo filing. Subjects in treatment were rolled over to the 20140159 study.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110100; 2011-004618-40 (EudraCT Number)
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Chronic Kidney Disease; Hyperparathyroidism, Secondary
Keywords: Dialysis; Sensipar; Mimpara; Hemodialysis; Peritoneal Dialysis; Renal; Parathyroid hormone; Pediatric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — Cinacalcet; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cinacalcet (Experimental): Prior to the partial clinical hold, the starting dose was 0.25 mg/kg (based on dry weight) and was titrated upwards (maximum allowed daily dose of 4.2 mg/kg) based on plasma intact parathyroid hormone (iPTH), corrected serum calcium levels obtained monthly, and adverse signs and symptoms.
  After the partial clinical hold the starting dose was 0.20 mg/kg (based on dry weight) and was titrated upwards (maximum allowed daily dose of 2.5 or 60 mg, whichever was lower) based on plasma iPTH, corrected serum calcium levels obtained monthly, weekly monitoring of ionized calcium levels, and adverse signs and symptoms.
  All participants also received standard of care, which may have included vitamin D sterols.
  Interventions: Drug: Cinacalcet hydrochloride; Drug: Standard of Care

INTERVENTIONS:
Drug: Cinacalcet hydrochloride — Cinacalcet was provided as 5 mg capsules that were opened, and the contents were either sprinkled on soft food or suspended into a sucrose syrup to create a liquid suspension for administration. All doses were administered with food or shortly after a meal at the same time daily.
  Other Names: Sensipar®; Mimpara®
Drug: Standard of Care — Standard of care may have included vitamin D sterols (25 OH vitamin D and/or 1-25 OH vitamin D and its analogs) at the discretion of the investigator.

SUMMARY:
The primary objective was to characterize corrected serum calcium levels on treatment with cinacalcet in pediatric patients with secondary hyperparathyroidism (HPT).

DETAILED DESCRIPTION:
This is a multicenter, 26-week, single-arm, open-label, safety study. Participants were to remain on study for 26 weeks or until time of kidney transplantation, whichever came first.

The study and enrollment was placed on partial clinical hold in February 2013 which resulted in changes to the protocol. The study was restarted in April 2014 following these changes.

Participants who completed the 26-week study or were on study when the study was closed in June 2016 were eligible to participate in an open-label extension study (Study 20140159; NCT02341417).

ELIGIBILITY:
Inclusion criteria:

* Subjects between the ages of 28 days to < 6 years of age at enrollment (Czech Republic minimum age is ≥ 2 years of age at enrollment)
* Screening plasma iPTH level > 300 pg/mL (31.8 pmol/L) from the central laboratory, and not have received any cinacalcet therapy for at least 30 days prior to start of dosing
* Screening corrected calcium from the central laboratory:
* ≥ 9.4 mg/dL (2.35 mmol/L) if age 28 days to < 2 years
* ≥ 8.8 (2.2 mmol/L) if age ≥ 2 to < 6 years
* Serum phosphorus from the central laboratory:
* ≥ 5.0 mg/dL (1.25 mmol/L) if age 28 days to < 1 year
* ≥ 4.5 mg/dL (1.13 mmol/L) if age ≥ 1 to < 6 years
* SHPT not due to vitamin D deficiency, per investigator assessment
* Dry weight ≥ 7 kg at the time of screening

Exclusion criterion:

* History of congenital long QT syndrome, second or third degree heart block, ventricular tachyarrhythmias or other conditions associated with prolonged QT interval
* Corrected QT interval (QTc) > 500 ms, using Bazett's formula
* QTc ≥ 450 to ≤ 500 ms, using Bazett's formula, unless written permission to enroll is provided by the investigator after consultation with a pediatric cardiologist
* Use of grapefruit juice, herbal medications, or potent CYP 3A4 inhibitors (e.g., erythromycin, clarithromycin, ketoconazole, itraconazole)
* Use of concomitant medications that may prolong the QTc interval (e.g., ondansetron, albuterol)

Ages: 28 Days to 2189 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2012-06-22 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- United States (17):
  - Research Site, Birmingham, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, The Bronx, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Research Site, Prague, Czechia
- France (3):
  - Research Site, Bron
  - Research Site, Lille
  - Research Site, Paris
- Research Site, Heidelberg, Germany
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
- Italy (3):
  - Research Site, Genova
  - Research Site, Roma
  - Research Site, Torino
- Research Site, Chihuahua City, Mexico
- Research Site, Amsterdam, Netherlands
- Research Site, Grafton, Auckland, New Zealand
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Košice, Slovakia

REFERENCES:
- [Background] Chen P, Sohn W, Narayanan A, Gisleskog PO, Melhem M. Bridging adults and paediatrics with secondary hyperparathyroidism receiving haemodialysis: a pharmacokinetic-pharmacodynamic analysis of cinacalcet. Br J Clin Pharmacol. 2019 Jun;85(6):1312-1325. doi: 10.1111/bcp.13900. Epub 2019 Apr 25. PMID 30756425
- [Background] Warady BA, Ng E, Bloss L, Mo M, Schaefer F, Bacchetta J. Cinacalcet studies in pediatric subjects with secondary hyperparathyroidism receiving dialysis. Pediatr Nephrol. 2020 Sep;35(9):1679-1697. doi: 10.1007/s00467-020-04516-4. Epub 2020 May 4. PMID 32367309
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 study centers in Czech Republic (1 site), France (1 site), Germany (1 site), Italy (1 site), Slovakia (1 site), Poland (3 sites), and the United States (6 sites). The first participant was enrolled on 22 June 2012, and the last participant completed the study on 03 June 2016.
Pre-assignment Details: Because of changes to the study design that were implemented after the partial clinical hold, data are presented overall and for 2 cohorts: participants enrolled before the partial clinical hold (Cohort 1) and participants enrolled after the partial clinical hold (Cohort 2).
Groups:
- Cohort 1: Cohort 1 consists of participants enrolled before the partial clinical hold. Participants received cinacalcet administered daily for 24 weeks. The starting dose was 0.25 mg/kg (based on dry weight) with dose adjustments and withholding based on plasma intact parathyroid hormone (iPTH), corrected serum calcium levels obtained monthly, and adverse signs and symptoms; the maximum allowed daily dose was 4.2 mg/kg.
- Cohort 2: Cohort 2 consists of participants enrolled after the partial clinical hold. Participants received cinacalcet administered daily for 24 weeks. The starting dose was 0.20 mg/kg (based on dry weight) with dose adjustments and withholding based on plasma iPTH, corrected serum calcium levels obtained monthly, weekly monitoring of ionized calcium levels, and adverse signs and symptoms; the maximum allowed daily dose was 2.5 mg/kg/day or 60 mg, whichever was lower.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 8 | 10
Received Treatment | 7 | 10
Completed | 2 | 2
Not Completed | 6 | 8
Not completed — Non-compliance | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Administrative Decision | 4 | 5
Not completed — Protocol-specified Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: months] | 37.1 (18.9) | 35.0 (15.9) | 35.9 (16.8)
Age, Customized [Number; unit: participants]
  28 days to < 2 years | 2 | 1 | 3
  2 years to < 6 years | 6 | 9 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 6 | 9 | 15
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 7 | 8 | 15
Corrected Serum Calcium [Mean (Standard Deviation); unit: mg/dL] | 10.56 (0.75) | 9.82 (0.61) | 10.15 (0.76)
Intact Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] | 1414.34 (699.90) | 1206.92 (597.85) | 1299.11 (634.18)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hypocalcemia
Description: Hypocalcemia was defined as corrected serum calcium levels < 9.0 mg/dL (2.25 mmol/L) for participants aged 28 days to < 2 years, and < 8.4 mg/dL (2.1 mmol/L) for participants aged ≥ 2 years to < 6 years at any time during the study.
Time Frame: 26 weeks
Population: The analysis included participants who received at least 1 dose of cinacalcet and had at least 1 measured serum calcium value while on cinacalcet (calcium analysis set).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Total: Participants received cinacalcet administered daily for 24 weeks.
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percentage of participants | 0.0 [0.0 to 34.8] | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 16.2]

2. Secondary Outcome: Percentage of Participants With Corrected Serum Calcium Levels < 8.8 mg/dL (2.2 mmol/L) During the Study
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percentage of participants | 14.3 [0.7 to 52.1] | 10.0 [0.5 to 39.4] | 11.8 [2.1 to 32.6]

3. Secondary Outcome: Percent Change From Baseline in Intact Parathyroid Hormone (iPTH)
Time Frame: Baseline and weeks 3, 7, 11, 15, 19, 22, and 24
Population: The analysis included all enrolled participants with at least 1 post-baseline assessment (full analysis set) and with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percent change
  Week 3 (n = 7, 9, 16) | -22.96 (64.67) | -3.37 (54.82) | -11.94 (58.11)
  Week 7 (n = 4, 9, 13) | 3.87 (110.94) | -3.13 (52.94) | -0.98 (70.40)
  Week 11 (n = 4, 8, 12) | -51.70 (27.18) | -7.15 (75.30) | -22.00 (65.51)
  Week 15 (n = 2, 7, 9) | -65.31 (6.83) | -51.69 (39.91) | -54.71 (35.16)
  Week 19 (n = 1, 3, 4) | -79.02 (NA) — Could not be calculated for a sample size = 1 | -57.35 (32.86) | -62.76 (28.93)
  Week 22 (n = 0, 1, 1) | NA (NA) — No participants with available data | -78.04 (NA) — Could not be calculated for a sample size = 1 | -78.04 (NA) — Could not be calculated for a sample size = 1
  Week 24 (n = 0, 1, 1) | NA (NA) — No participants with available data | -67.42 (NA) — Could not be calculated for a sample size = 1 | -67.42 (NA) — Could not be calculated for a sample size = 1

4. Secondary Outcome: Percent Change From Baseline in Corrected Serum Calcium
Time Frame: Baseline and weeks 3, 7, 11, 15, 19, 22, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percent change
  Week 3 (n = 7, 10, 17) | -0.50 (4.47) | 3.43 (6.38) | 1.81 (5.86)
  Week 7 (n = 4, 8, 12) | -3.58 (12.23) | 3.60 (9.31) | 1.21 (10.41)
  Week 11 (n = 4, 8, 12) | -3.23 (10.51) | 1.46 (5.24) | -0.10 (7.28)
  Week 15 (n = 2, 7, 9) | -6.86 (12.44) | 2.99 (5.09) | 0.80 (7.59)
  Week 19 (n = 1, 3, 4) | 1.94 (NA) — Could not be calculated for a sample size of 1 | -0.49 (6.62) | 0.12 (5.54)
  Week 22 (n = 0, 1, 1) | NA (NA) — No participants with available data | 5.88 (NA) — Could not be calculated for a sample size of 1 | 5.88 (NA) — Could not be calculated for a sample size of 1
  Week 24 (n = 0, 1, 1) | NA (NA) — No participants with available data | 2.94 (NA) — Could not be calculated for a sample size of 1 | 2.94 (NA) — Could not be calculated for a sample size of 1

5. Secondary Outcome: Percent Change From Baseline in Serum Phosphorous
Time Frame: Baseline and weeks 3, 7, 11, 15, 19, 22, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percent change
  Week 3 (n = 7, 10, 17) | -10.75 (32.49) | -5.11 (39.32) | -7.43 (35.69)
  Week 7 (n = 4, 8, 12) | -8.68 (20.88) | -9.60 (29.79) | -9.29 (26.15)
  Week 11 (n = 4, 8, 12) | 14.39 (22.18) | 4.54 (39.08) | 7.82 (33.61)
  Week 15 (n = 2, 7, 9) | 13.99 (26.33) | -16.07 (28.14) | -9.39 (29.26)
  Week 19 (n = 1, 2, 3) | 10.87 (NA) — Could not be calculated for sample size of 1 | 3.45 (4.88) | 5.92 (5.50)
  Week 22 (n = 0, 1, 1) | NA (NA) — No participants with available data | -1.72 (NA) — Could not be calculated for a sample size of 1 | -1.72 (NA) — Could not be calculated for a sample size of 1
  Week 24 (n = 0, 1, 1) | NA (NA) — No participants with available data | 8.62 (NA) — Could not be calculated for a sample size of 1 | 8.62 (NA) — Could not be calculated for a sample size of 1

6. Secondary Outcome: Percent Change From Baseline in Calcium Phosphorus Product (Ca x P)
Time Frame: Baseline and weeks 3, 7, 11, 15, 19, 22, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percent change
  Week 3 (n = 7, 10, 17) | -1.89 (39.00) | -2.72 (38.08) | -2.37 (37.23)
  Week 7 (n = 4, 8, 12) | -11.56 (26.35) | -6.83 (29.97) | -8.40 (27.68)
  Week 11 (n = 4, 8, 12) | 9.48 (17.84) | 5.74 (38.78) | 6.99 (32.36)
  Week 15 (n = 2, 7, 9) | 7.58 (38.39) | -14.24 (28.24) | -9.39 (29.58)
  Week 19 (n = 1, 2, 3) | 12.34 (NA) — Could not be calculated for a sample size of 1 | 6.41 (9.06) | 8.39 (7.27)
  Week 22 (n = 0, 1, 1) | NA (NA) — No participants with available data | 3.37 (NA) — Could not be calculated for a sample size of 1 | 3.37 (NA) — Could not be calculated for a sample size of 1
  Week 24 (n = 0, 1, 1) | NA (NA) — No participants with available data | 10.96 (NA) — Could not be calculated for a sample size of 1 | 10.96 (NA) — Could not be calculated for a sample size of 1

7. Secondary Outcome: Percentage of Participants Who Achieved > 30% Reduction in iPTH From Baseline at Any Two Consecutive Measurements
Description: A participant was considered to have achieved > 30% reduction in iPTH from baseline at any 2 consecutive measurements if percent change of any two consecutive post-baseline iPTH values were < -30% regardless if there was a missing value in between.
Time Frame: 26 weeks
Population: The analysis included all enrolled participants with at least 1 post-baseline assessment (full analysis set).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percentage of participants | 57.1 [22.5 to 87.1] | 40.0 [15.0 to 69.6] | 47.1 [26.0 to 68.9]

8. Secondary Outcome: Percentage of Participants Who Achieved ≥ 30% Reduction in iPTH From Baseline During the Study
Description: A participant was considered to have achieved ≥ 30% reduction in iPTH if the percent change of any post-baseline iPTH value was ≤ -30% from baseline.
Time Frame: 26 weeks
Population: The analysis included all enrolled participants with at least 1 post-baseline assessment (full analysis set).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percentage of participants | 100.0 [65.2 to 100.0] | 50.0 [22.2 to 77.8] | 70.6 [47.8 to 87.6]

9. Secondary Outcome: Percentage of Participants Who Achieved iPTH Values Between 200 and 300 pg/mL at Any Two Consecutive Measurements
Description: A participant was considered to have achieved iPTH between 200 and 300 pg/mL (21.2 and 31.8 pmol/L) at any 2 consecutive measurements if any two consecutive post-baseline iPTH values were within the range regardless if there was a missing value in between. The analysis included all enrolled subjects with at least 1 post-baseline assessment.
Time Frame: 26 weeks
Population: The analysis included all enrolled participants with at least 1 post-baseline assessment (full analysis set).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percentage of participants | 0.0 [0.0 to 34.8] | 10.0 [0.5 to 39.4] | 5.9 [0.3 to 25.0]

10. Secondary Outcome: Percentage of Participants Who Achieved iPTH Values < 300 pg/mL During the Study
Description: A participant was considered to have achieved iPTH < 300 pg/mL (31.8 pmol/L) during the study if any post-baseline iPTH value was < 300 pg/mL.
Time Frame: 26 weeks
Population: The analysis included all enrolled subjects with at least 1 post-baseline assessment (full analysis set).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 7 | 10 | 17
percentage of participants | 57.1 [22.5 to 87.1] | 50.0 [22.2 to 77.8] | 52.9 [31.1 to 74.0]

11. Secondary Outcome: Dose- and Weight-Normalized Maximum Plasma Concentration (Cmax) of Cinacalcet
Time Frame: Week 12
Population: The Pharmacokinetic/ Pharmacodynamic (PK/PD) analysis set includes all participants who received at least one dose of study drug and had at least one evaluable PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL/(mgkg)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 7
ng/mL/(mgkg) | 15.1 (16.6) | 17.8 (10.0)

12. Secondary Outcome: Dose- and Weight-Normalized Area Under the Plasma Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUClast) for Cinacalcet
Time Frame: Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hr*ng/mL/(mgkg)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 6
hr*ng/mL/(mgkg) | 160 (195) | 176.8 (177)

ADVERSE EVENTS:
Time Frame: 26 Weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Cohort 1 | Cohort 2 | Total
Serious Adverse Events (participants affected / at risk) | 4/7 | 5/10 | 9/17
Other Adverse Events (participants affected / at risk) | 5/7 | 9/10 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=10) | Total (N=17)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Complication associated with device (General disorders) | 1 | 1 | 2
Adenovirus infection (Infections and infestations) | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Device related sepsis (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Device malfunction (Product Issues) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=10) | Total (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 4
Asthenia (General disorders) | 0 | 1 | 1
Complication associated with device (General disorders) | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 2 | 3
Bronchitis (Infections and infestations) | 2 | 0 | 2
Device related sepsis (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4
Viral infection (Infections and infestations) | 2 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Catheter removal (Surgical and medical procedures) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.